CLINICAL TRIAL: NCT01244243
Title: Robot-Assisted Hand Motor Therapy for Subjects With Hemiparetic Stroke
Acronym: Robot3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS#2004-3852
Record Dates: First submitted 2010-11-03; First posted 2010-11-19 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: stroke; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active therapy (Experimental): All subjects receive the same active robotic therapy, there is no placebo arm, as a key goal of this study is to define predictors of response to active treatment.
  Interventions: Device: Hand & Wrist Assisting Robotic Device

INTERVENTIONS:
Device: Hand & Wrist Assisting Robotic Device — Treatment occurs in 2 hour sessions, 4 times a week over 3 weeks. In each treatment session, you will sit in a chair and have your weak hand attached to a mechanical device (the robot), which will help you open and close your hand. During the treatment, different types of objects (with varying shapes, sizes, and weight) will be placed into your hand. You will be given a variety of instructions related to the grasping, feeling, or identifying of the object in your hand. Sometimes these instructions will be given from the investigator and sometimes from the computer. You will often be asked to grasp, or release, each of these objects as best you can. You will also be asked to concentrate on the object in your hand. An example of what you may be asked to do is to name the object. During other times, you will play games, using the robot to control game parts on the computer screen. At other times, you will move your hand so that the robot can measure your hand function.
  Other Names: HWARD

SUMMARY:
The purpose of this study is to develop and assess the effectiveness of robot-assisted movement therapy in enhancing hand motor function in subjects with chronic hemiparetic stroke, and to identify predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Had stroke between 11-26 weeks ago
3. Have some weakness in one of your wrists or hands due to stroke
4. Did not have too much disability prior to stroke
5. Do not have major depression

Exclusion Criteria:

1. Non-English speaking
2. If you have trouble keeping good attention
3. Pregnant, advanced liver, kidney, heart, or lung disease
4. Terminal medical diagnosis or major neurological or psychiatric disease apart from stroke
5. Cannot undergo MRI scanning
6. Have history of brain surgery or seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Cramer, MD, Principal Investigator — University of Californai Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Derived] McKenzie A, Dodakian L, See J, Le V, Quinlan EB, Bridgford C, Head D, Han VL, Cramer SC. Validity of Robot-Based Assessments of Upper Extremity Function. Arch Phys Med Rehabil. 2017 Oct;98(10):1969-1976.e2. doi: 10.1016/j.apmr.2017.02.033. Epub 2017 May 5. PMID 28483654

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Therapy
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Therapy: All subjects receive the same active robotic therapy, there is no placebo arm, as a key goal of this study is to define predictors of response to active treatment.
  Hand & Wrist Assisting Robotic Device: Treatment occurs in 2 hour sessions, 4 times a week over 3 weeks.
Arm/Group | Active Therapy
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test
Description: The Action Research Arm Test is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from: 3: Performs test normally 2: Completes test, but takes abnormally long or has great difficulty 1: Performs test partially 0: Can perform no part of test. The test is used to determine upper limb function, 0-57 points with higher is better, 57 is the highest score indicating normal arm movement.
Time Frame: change from baseline to 1 month post-end treatment, Intention To Treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Therapy
Number analyzed (Participants) | 41
units on a scale | 4.1 [2.3 to 5.9]

2. Primary Outcome: Arm Motor Fugl-Meyer Test
Description: The Arm Motor Fugl-Meyer test is an assessment of Sensorimotor Recovery After Stroke. It is a 33 item measure with 3 subgroups which are Proximal, Wrist/Hand, and Coordination/Speed. The scaling for each item works on a scale of 0-2 with 0 being not able to be done, 1 being partially done, and 2 being done normally. The scoring goes from 0-66, higher is better, 66 is considered a normal score with no noticable complications in movement.
Time Frame: change from baseline to 1 month post-end treatment, Intention To Treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Therapy
Number analyzed (Participants) | 41
units on a scale | 3.7 [2.7 to 4.8]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Active Therapy
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No